CLINICAL TRIAL: NCT04746651
Title: Evaluating the Feasibility of a Guided Self-help Programme for an Adult Male Population of Offenders Serving a Long-term Prison Sentence
Brief Title: A Feasibility Study of a Guided Self-help Programme for Male Offenders Serving a Long-term Prison Sentence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Lanarkshire (Other Government)
Responsible Party: Principal Investigator, Jennifer Lai, Trainee Clinical Psychologist, University of Glasgow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L19007
Record Dates: First submitted 2019-02-11; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Anxiety; Depression
Keywords: Feasibility study; Prisoners; Male offenders; Guided self help; Anxiety; Low mood
MeSH Terms: conditions — Anxiety Disorders; Depression; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Self Help (Experimental): Four guided self-help booklets were used; "Why do I feel so bad?" covered formulation/understanding feelings, "I can't be bothered doing anything" centred on activity scheduling, "Why does everything always go wrong?" focused on thought-challenging, and "How to fix almost everything" incorporated problem solving. Linked worksheets were adapted following feedback from Prison Officers.
  Interventions: Other: Guided Self Help

INTERVENTIONS:
Other: Guided Self Help — Guided self help appointments with prison staff - 4x 30 minute appointments.

SUMMARY:
Background: Prisoners have complex mental health needs, and there is a disproportionately higher incidence of mental health problems compared with the general population. Although research indicates that psychological interventions are effective in treating prisoners with anxiety and depression, medication is often the only treatment available in prisons. Living Life To The Full (LLTTF) is a life skills programme teaching skills to cope with life stresses, and has been shown to reduce anxiety and depression in individuals in the community.

Research Questions

1. Will prisoners take part in and engage with LLTTF?
2. Do LLTTF booklets need to be adapted for prisoners?
3. Does LLTTF show an effect of reducing anxiety and/or depression?
4. Does history of HI reduce responsivity to LLTTF?
5. Does LLTTF reduce number of breaches of prison rules?

What did the study involve?: Prison Officers in HMP Shotts were invited to take part and attend LLTTF training. Male prisoners aged 21 and above in HMP Shotts were recruited using posters. Assessment of anxiety, depression, perceived functioning, and history of head injury was carried out. Prisoners' work attendance and breaches of prison rules for the month prior to and month during LLTTF was collected. Prison Officers and prisoners provided feedback of LLTTF at end of treatment.

Results: Six (6%) Prison Officers attended LLTTF training and two (33%) withdrew prior to prisoner recruitment. 6% (n=15) of prisoners invited to take part volunteered and were eligible. Seven prisoners completed LLTTF.

There was a sign of a treatment effect with reductions in depression following LLTTF. Anxiety reduced at the last session and increased at post-treatment, which reflects the deterioration in a minority of prisoners. Due to the small sample size, history of HI and responsivity was not explored. Prisoners were not on report the month prior to LLTTF, therefore impact on breached rules was not explored.

Feedback from Prison Officers and prisoners indicated materials required adaptation for prison, such as including activities feasible in prison. Prison Officers highlighted practical barriers to delivery of LLTTF, including limited time.

Conclusions: Guided self-help in prison is worth pursuing. Revision of materials with Prison Officers and prisoners is recommended, and evaluated in future research. Due to practical barriers reported by Prison Officers, designated guided self-help workers may be better placed to deliver this intervention.

ELIGIBILITY:
Eligible prisoners were adult males (aged 21+) at HMP Shotts who experienced mild-severe levels of psychological distress (defined as PHQ score of 5+), were prepared to attend four sessions of the guided self-help, able to read and write, and able to engage in the guided self-help.

Prisoners were excluded if deemed, by Prison Officers or healthcare staff, to pose a direct risk of harm to the field researcher (or were at risk of imminent and significant self-harm).

Ages: 21 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
The number of prison officers who complete the LLTTF training and the number of prisoners who complete the 4 appointments of LLTTF. | Through study completion, 17/01/2020
  Quantitative

SECONDARY OUTCOMES:
Reports of the means of the PHQ-9 | Through study completion, an average of 4 weeks for each participant.
  Quantitative
Reports of the means of the GAD-7 | Through study completion, average of 4 weeks for each participant.
  Quantitative
The percentage of participants who believe the booklets need to be adapted for use in prison. | Through study completion, 17/01/2020
  Quantitative

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom